CLINICAL TRIAL: NCT01745276
Title: Evaluation of Bisphosphonate Coated Pins for Extern Fixation in Tibia Osteotomy
Acronym: PFX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Addbio AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: PFX-2009378
Record Dates: First submitted 2012-05-23; First posted 2012-12-10 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Osteoarthritis
Keywords: Pin fixation; Osteotomy; hemicallotasis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- External pins coated by biphosfonate. (Experimental): External pins coated by biphosfonate.
  Interventions: Device: Biphosfonate
- External pins coated by hydroxylapatite. (Active Comparator): External pins coated by hydroxylapatite.
  Interventions: Device: Hydroxylapatit

INTERVENTIONS:
Device: Biphosfonate — External pins coated by biphosfonate.
  Arms: External pins coated by biphosfonate.
Device: Hydroxylapatit — External pins coated by Hydroxylapatit.
  Arms: External pins coated by hydroxylapatite.

SUMMARY:
The purpose of this study is to evaluate the relative osseomechanical strength of a novel coated pin/screw in a clinical model.

DETAILED DESCRIPTION:
The pin fixation and the risk for pin loosening and pintract infection is intimately connected Moroni et al., Magyar et al. Toksvig-Larsen and W-Dahl) The pin performance ratio for insertion to extraction torque (PPI) varies significantly between screw types.

The extraction torque force is the most important value and it is estimated that a removal torque around 300 Nm probably will be the best bon-pin fixation in clinical practice.

In animal studies and even in clinical studies the hydroxyapatite (HA) coated screw retained the highest level of osseointegration. However, the fixation for HAscrews is, especially in diaphyseal bone, the risk for too tight fixation, with extreme difficulties to remove the screws in few cases as a result ( high pain and seldom it is impossible to remove the screw) Coating by biphosphonate is a new novel technique with preclinical appealing performance, which theoretically should make this coating very appealing in clinical practice. The theory behind this technique is that it create a good pinfixation reasonable easy to remove.

The current most used cortical screw designs performed poorest in terms of fixation (PPI)

Method

Using the hemicallotasis technique for correction in high tibial osteotomies today, HA coated (Osteotite) conical 130/50 screws is used in the proximal tibia - the metaphysic - and plain (standard) cortical conical screws 110/40 is used in the diaphysis.

To study the effect of an improved pin coating a study including 30 patients randomised to the standard procedure today or the novel technique using biphosphonate coated screws.

In the metaphysic, the randomisation will be between the HA coated (Osteotite) screws and the biphosphonated coated screws 130/50 (screw thread 50mm) In the diaphysis the randomisation will be between the plain standard 110/40 screws and the biphosphonate 110/40 coated screws

Totally 30 patients will be studied which means totally 120 pins. This has been based on power calculations resulting in 23 patients in each group and calculated on extraction torque force. This is a clinical study and 30 patients is estimated due to expected drop out.

ELIGIBILITY:
Inclusion Criteria:

* All patients which are diagnosed with arthr and needs an operation.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the relative osseomechanical strength of a novel coated pin/screw in a clinical mode. | 2011-07-01-2012-02-01
  To evaluate the relative osseomechanical strength of a novel coated pin/screw

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopeadic Clinic Hospital, Hässleholm, Sweden